# BIOEQUIVALENCE STUDY PROTOCOL

BIOEQUIVALENCE STUDY OF ACYCLOVIR 200 MG TABLET MANUFACTURED BY PT. KIMIA FARMA (PERSERO) TBK IN COMPARISON WITH ZOVIRAX® 200 MG TABLET MANUFACTURED BY GLAXO WELLCOME S.A., ARANDA, SPAIN, PACKED BY GLAXOSMITHKLINE AUSTRALIA PTY LTD, BORONIA, AUSTRALIA, IMPORTED BY PT. GLAXO WELLCOME INDONESIA, JAKARTA, INDONESIA

Protocol No.: 515/STD/PML/2019

**Drug Substance** 

Acyclovir 200 mg

**Sponsor** 

PT. Kimia Farma (Persero) Tbk

Jl. Rawa Gelam V No. 1

Jakarta, Indonesia

Tel

: +62 21 4609354

Fax

: +62 21 4603143

**Study Centre** 

PT. Pharma Metric Labs

Gedung Indra Sentral Cempaka Putih Unit R-U

Jalan Letjen Suprapto Kav. 60

Central Jakarta, 10520

Indonesia

Tel: +62 21 4265310

Fax: +62 21 4210302

**Principal Investigator** 

Metta Sinta Sari Wiria, Pharm, MS

**Study Director** 

I Gusti Putu Bagus Diana Virgo, Pharm

**Protocol Author** 

Olivia Valencia, Pharm

Issue date

13 December 2019

Version

00

Confidentiality Statement

The confidential information in this document is provided to the sponsor for review. The sponsor acceptance of this document constitutes agreement that the sponsor will not disclose the information herein to others without written authorization from the Principal Investigator and PT. Pharma Metric Labs. Do not copy this protocol without written permission from the Principal Investigator and PT. Pharma Metric Labs.

## 

#### 1. TITLE PAGE

#### 1.1. Study Title

Bioequivalence study of Acyclovir 200 mg tablet manufactured by PT. Kimia Farma (Persero) Tbk in comparison with Zovirax 200 mg tablet manufactured by Glaxo Wellcome S.A., Aranda, Spain, Packed by GlaxoSmithKline Australia Pty Ltd, Boronia Australia, imported by PT. Glaxo Wellcome Indonesia, Jakarta, Indonesia.

## 1.2. Name, person in charge and address of Sponsor

Dra. Dyah Juliana Pudjiati, M.Kes., Apt Regulatory Affairs PT. Kimia Farma Tbk Jl Veteran No. 9 Jakarta 11010 Telp. (62-21) - 3847709 Fax. (62-21) - 3814441

## 1.3. Name, person in charge and address of Institution

I Gusti Putu Bagus Diana Virgo, Pharm PT. Pharma Metric Labs Gedung Indra Sentral Cempaka Putih Unit R-U Jalan Letjen Suprapto Kav. 60 Central Jakarta, 10520 Indonesia

Tel : +62 21 4265310 Fax : +62 21 4210302

Email: gusti.virgo@pharmametriclabs.com

## 1.4. Name and address of Principal Investigator

Metta Sinta Sari Wiria, Pharm, MS University of Indonesia Jalan Salemba Raya No.6, Jakarta Pusat Jakarta 10430

#### 1.5. Name of Study Physician

Jessica, MD, SpOk

#### 1.6. Name and address of clinical laboratory

Tri Handayani Pramita Clinical Laboratory Jalan Matraman Raya, No. 26, East Jakarta, Indonesia. Tel: +62 21 85908530

Tel: +62 21 85908530 Fax: +62 21 8502039

515/STD/PML/2019

# 

#### 1.7. Name, person in charge and address of analytical laboratory

Seriyati Naibaho, Chem

PT. Pharma Metric Labs

Gedung Indra Sentral Cempaka Putih Unit R-U

Jalan Letjen Suprapto Kav. 60

Central Jakarta, 10520

Indonesia

Tel : +62 21 4265310 Fax : +62 21 4210302

# 1.8. Name, person in charge and address for pharmacokinetics and statistical analysis

Niken Pratiwi, Pharm

PT. Pharma Metric Labs

Gedung Indra Sentral Cempaka Putih Unit R-U

Jalan Letjen Suprapto Kav. 60

Central Jakarta, 10520

Indonesia

Tel : +62 21 4265310

Fax : +62 21 4210302

# 1.9. Name of other study personnel

Study Director : I Gusti Putu Bagus Diana Virgo, Pharm

Clinical : Uluk Suharsi Putra, Chem

Quality Assurance : Hanoum Kayasa Swasti, Chem. Eng

### 1.10. Start and end date of clinical and analytical study

Dates of Clinical Portion:

Screening : After protocol approval from NADFC

Period 1 : After completion of screening process

Period 2 : One week after Period 1

Dates of Analytical Portion:

Method Validation : January 2016

Sample Analysis : After completion of Period 2

## INVESTIGATOR SIGNATURE PAGE

The undersigned hereby confirmed that the protocol had been read and understood, and agreed to abide by the procedures as stipulated. We agreed to conduct the study with reference to The Indonesian Good Clinical Practice Guideline 2016; The Indonesian Bioequivalence Study Guideline BPOM 2015; ASEAN Guidelines for The Conduct of Bioavailability and Bioequivalence Study 2015; EMA Guideline on the Investigation of Bioequivalence 2010; USFDA Guidance for Industry on Bioavailability and Bioequivalence Studies for Orally Administered Drug Products 2003; Declaration of Helsinki and the International Conference on Harmonization Good Clinical Practice Guideline.

| Responsibility | Name | Signature and date |
|---|---|---|
| Principal Investigator | Metta Sinta Sari Wiria, Pharm, MS | Mel 67 DAN 2020 |
| Study Director | I Gusti Putu Bagus Diana Virgo, Pharm | O3 Jan 2020 |
| Study Physician | Hendi Tri Ariatmoko, MD | Of money |
| Clinical | Uluk Suharsi Putra, Chem | CPOP 08 VAN 2020 |
| Analytical | Seriyati Naibaho, Chem | 06 Jan 2019 00 Jan 202 |
| Quality Assurance | Hanoum Kayasa Swasti, Chem.Eng | Hanoust C Jan 2020 |
| Statistician | Niken Pratiwi, Pharm | MAP 08 Jan 2020 |
| Sponsor | Dra. Dyah Juliana Pudjiati, M.kes., Apt | Mars 09/200 2000 |

# 2. PROTOCOL SYNOPSIS

| Title of Study | Bioequivalence study of Acyclovir 200 mg tablet manufactured by PT. Kimia Farma (Persero) Tbk in comparison with Zovirax <sup>®</sup> 200 mg tablet manufactured by Glaxo Wellcome S.A., Aranda, Spain, Packed by GlaxoSmithKline Australia Pty Ltd, Boronia Australia, imported by PT. Glaxo Wellcome Indonesia, Jakarta, Indonesia. |
|---|---|
| Objectives | The objective of this study is to investigate whether Acyclovir 200 mg tablet manufactured by PT. Kimia Farma (Persero) Tbk is bioequivalent to its reference product, Zovirax® 200 mg tablet manufactured by Glaxo Wellcome S.A., Aranda, Spain, Packed by GlaxoSmithKline Australia Pty Ltd, Boronia Australia, imported by PT. Glaxo Wellcome Indonesia, Jakarta, Indonesia. |
| Study Design | Randomized, single-blind, single-dose, 2-period, 2-treatment, 2-sequence, 2-way crossover study in healthy subjects under fasting condition. |
| Number of<br>Subjects | 28 healthy subjects |
| Washout period | 1 week between each treatment |
| · | Name : Acyclovir 200 mg tablet |
| | Manufacturer : PT. Kimia Farma (Persero) Tbk |
| | Reg No : GKL9812415010A1 |
| Test Product | Batch No : C90576J |
| | Mfg Date : March 2019 |
| | Exp Date : March 2024 |
| Reference Product | Name : Zovirax® 200 mg tablet |
| | Manufacturer : Glaxo Wellcome S.A., Aranda, Spain, Packed by Glaxo-<br>SmithKline Australia Pty Ltd, Boronia Australia, imported<br>by PT. Glaxo Wellcome Indonesia, Jakarta, Indonesia. |
| | Reg No : DKI1691601310A1 |
| | Batch No : 243E |
| | Mfg Date : March 2018 |
| | Exp Date : March 2020 |
| Inclusion Criteria | <ul> <li>have read the subject information and signed informed consent documents</li> <li>healthy male and female</li> <li>age 18 – 55 years</li> <li>body mass index between 18–25 kg/m²</li> <li>have a normal electrocardiogram</li> <li>blood pressure within normal range (systolic 90-120 mmHg and diastolic 60-80 mmHg)</li> <li>heart rate within normal range (60-100 bpm)</li> <li>absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening</li> </ul> |

Date: 13 December 2019

515/STD/PML/2019

# Pharma∬\etric Labs

| | 1 |
|---|---|
| Exclusion Criteria | <ul> <li>pregnant and/or nursing women</li> <li>history of contraindication or hypersensitivity to acyclovir, or other antiviral or other ingredients in the study products or a history of serious allergic reaction to any drug, a significant allergic disease, or allergic reaction</li> <li>history or presence of medical condition which might significantly influence the pharmacokinetic of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.</li> <li>history or presence of any coagulation disorder or clinically significant hematology abnormalities</li> <li>using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day</li> <li>have participated in any clinical study within 3 months prior to the study (&lt; 90 days)</li> <li>have donated or lost 300 ml (or more) of blood within 3 months prior to the study</li> <li>smoke more than 10 cigarettes a day</li> <li>positive to HIV, HBsAg, and HCV tests (to be kept confidential)</li> <li>history of drug or alcohol abuse within 12 months prior to screening for this study</li> <li>unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access</li> </ul> |
| Screening | Medical history, physical examination, laboratory tests (routine hematology, blood biochemistry and urinalysis), electrocardiograph, pregnancy test and HIV, HBsAg, and HCV tests are carried out to screen the subjects and to obtain eligible subjects who meet the inclusion and exclusion criteria. |
| Subjects' Restriction | <ul> <li>Abstain from taking any medication at least one week before and during study period (unless necessary)</li> <li>Not permitted to smoke, consume alcohol, milk, beverages or food containing xanthines (e.g., tea, coffee, chocolate) or fruit juice 24 hours prior and during study period</li> <li>Instructed to avoid severe physical exertion during sampling hours</li> </ul> |
| Standardization of study condition | <ul> <li>Subjects are instructed to stay one night before and during the sampling period</li> <li>Subjects are instructed to fast from 8 hours before until 4 hours after drug administration</li> <li>The menu served and meal taken by subjects are standardized and recorded</li> <li>Water can be consumed as desired except during the period of 1 hour before until 2 hours after drug administration</li> </ul> |

| Investigational Product Administration | A single dose of 200 mg acyclovir of the test drug or 200 mg acyclovir of the reference drug (according to randomization code) will be given orally to the subjects in sitting posture. The drug will be administered with 240 mL water. |
|---|---|
| Sampling Schedule | Blood samples for acyclovir assay (approximately 6 mL) are drawn into tubes containing anticoagulant (EDTA) before dosing (0 h) and at 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after dosing. The pre-dose sample (0 h) is collected within an hour before the first drug dosing SN01. |
| | A total volume of 192 mL of blood will be collected from each subject (2 periods x 16 sampling points x 6 mL per sampling point), 96 mL per period. This volume of blood will be used for pharmacokinetic analysis. |
| Subject Monitoring | Vital signs (blood pressure, pulse, respiration rate and body temperature) are monitored and recorded prior to drug administration, and subsequently at 1, 3, 6, 10, 12, and 24 hours after drug administration. |
| | The subjects' safety is monitored during the entire study under direct supervision by Study Physician at the study site. |
| Washout period | One week between each treatment |
| Analyte | Acyclovir concentration will be measured in plasma by a validated LC-MS/MS method. The LLoQ is 7.5 ng/mL for acyclovir. |
| Pharmacokinetics<br>Parameter | C <sub>max</sub> , AUC <sub>t</sub> , AUC <sub>inf</sub> , t <sub>max</sub> and t <sub>1/2</sub> will be determined. |
| Statistical Analysis | Bioequivalence of the two formulations will be assessed by comparing the AUC <sub>t</sub> and C <sub>max</sub> of acyclovir values after ln transformation of the concentration data. The geometric mean ratios (test/reference) of the ln-transformed data and their 90% confidence intervals will be further analyzed with a parametric method (analysis of variance/ANOVA) using Equiv Test <sup>®</sup> version 2.0 (Statistical Solution Ltd., Saugus. MA, USA) or manual calculation which has been validated to Equiv Test <sup>®</sup> . |
| Bioequivalence<br>Criteria | The two products are considered bioequivalent when the 90% confidence intervals of the acyclovir geometric mean ratio between test and reference products fall within the range of $80.00\text{-}125.00\%$ for AUC, and C <sub>max</sub> . |

515/STD/PML/2019 PT. Kimia Farma (Persero) Tbk Date: 13 December 2019 Version: 00 Page 7 of 25